CLINICAL TRIAL: NCT00033774
Title: Peripheral Blood Stem Cell Collection From Adult Volunteers
Brief Title: Stem Cell Collection for Adult Volunteers
Status: Terminated | Type: Observational
Why Stopped: There is another active NHLBI protocol for the collection of stem cells for research from healthy volunteers and no need for this separate Protocol.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020160; 02-H-0160
Record Dates: First submitted 2002-04-09; First posted 2002-04-10 (Estimated); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Sickle Cell
Keywords: Leukapheresis; G-CSF; Mobilization; Stem Cells; Adult; Natural History; Healthy Volunteer; HV; Normal Control

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — stem cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Eligible healthy volunteers 18 and older

SUMMARY:
This study will examine the development of stem cells (very immature cells produced by the bone marrow) and their potential to change into cells of other organ types. These cells will be studied for their potential use in creating replacement tissue for diseases ranging from diabetes to Parkinson s.

Healthy volunteers 18 years of age or older may be eligible for this study. Candidates will be screened with a medical history, physical examination, and blood tests.

Participants will undergo a process called 'stem cell mobilization and apheresis' to collect bone marrow stem cells. For five days before the collection they will receive injections of a hormone called G-CSF, which stimulates release of stem cells from the bone marrow into the bloodstream. On the fifth day of the injections, stem cells will be collected through apheresis. For this procedure, blood is collected through a catheter (plastic tube) placed in an arm vein and directed into a cell separator machine. There, the white cells and stem cells are separated from the other blood components through a spinning process and collected in a bag inside the machine. The rest of the blood is returned to the donor through a catheter in the other arm.

DETAILED DESCRIPTION:
The renewal of various tissues and organs at steady state or following damage relies upon a small population of locally residing tissue specific "stem cells" Stem cells from adult bone marrow represent an ideal stem cell source based on their ease of collection. In order to begin to explore the potential of adult bone marrow for the correction of genetic diseases that affect the blood such as sickle cell disease, we propose in vitro and in vivo mouse studies to examine the regulation of normal differentiation of hematopoietic stem cells collected from adult volunteers. In order to obtain adult hematopoietic stem cells in large numbers for in vitro and in vivo studies, volunteers will undergo mobilization with G-CSF for 5 consecutive days followed by large volume apheresis on the 5th day of G-CSF injection. The harvested product will be immunomagnetically purified for the primitive progenitor population and viably cryopreserved in multiple aliquots.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 or greater.

Normal renal function: creatinine less than1.5 mg/dL, proteinuria less than1+.

Normal liver function: bilirubin less than 2.5 mg/dL, ALT less than 2.5 times the upper limit of normal, all other transminases less than 2.5 times the upper limit of normal.

Normal blood counts: WBC 3,000-10,000/mm3, granulocytes greater than 1,500/mm3, platelets greater than 150,000/mm3, hemoglobin greater than 12.5g/dL, MCV within normal limits.

Female volunteers of childbearing age should have a negative serum pregnancy test within one week of beginning G-CSF administration.

Meets NIH Department of Transfusion Medicine (DTM) eligibility criteria for blood component donation for in vitro research use (negative serologic tests for syphilis, hepatitis B and C, HIV, and HTLV-1).

Ability to give informed consent to participate in the protocol.

EXCLUSION CRITERIA:

Any underlying hematologic disorder including sickle cell disease.

Active viral, bacterial, fungal, or parasitic infection.

History of autoimmune disease, such as rheumatoid arthritis or systemic lupus erythematosus.

History of cancer excluding squamous carcinoma of the skin and cervical carcinoma in situ.

History of cardiovascular disease or related symptoms such as chest pain or shortness of breath.

Any positive serum screening test as listed below.

Allergy to G-CSF or bacterial E. coli products.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will occur from a pool of normal volunteers. Volunteers who are not undergoing pretreatment with G-CSF will receive two hundred and fifty (250) dollars for the leukapheresis. Volunteers who undergo pretreatment with G-CSF will receive a payment of five hundred (500) dollars upon completion of 5 days of G-CSF, blood draws, and the leukapheresis. In the event of early withdrawal from the study before the leukapheresis, the volunteer will receive fifty (50) dollars for each visit to the hospital which includes blood draws and G-CSF administration.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2002-04-29 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Collection of peripheral blood stem cells via standard leukapheresis | 5 days
  To explore the control of normal differentiation of adult hematopoietic stem cells collected from the peripheral blood after G-CSF mobilization.

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wei G, Schubiger G, Harder F, Muller AM. Stem cell plasticity in mammals and transdetermination in Drosophila: common themes? Stem Cells. 2000;18(6):409-14. doi: 10.1634/stemcells.18-6-409. PMID 11072028
- [Background] Orkin SH. Diversification of haematopoietic stem cells to specific lineages. Nat Rev Genet. 2000 Oct;1(1):57-64. doi: 10.1038/35049577. PMID 11262875
- [Background] Lemischka I. Stem cell dogmas in the genomics era. Rev Clin Exp Hematol. 2001 Mar;5(1):15-25. doi: 10.1046/j.1468-0734.2001.00030.x. PMID 11486729
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2002-H-0160.html